CLINICAL TRIAL: NCT05894629
Title: Effects of an Active Coping Program in Patients With Persistent Post-Covid Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Laura Barrero Santiago, Phd Candidate, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LGCOVIDTRIAL
Record Dates: First submitted 2023-06-06; First posted 2023-06-08 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Long COVID; Pain
Keywords: Intervention; Long Covid Pain; Pain Neuroscience Education; Exercise
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Neuroscience Education (PNE)+ Therapeutic Exercise (TE) (Experimental): Intervention Group (IG):
  12-week program consisting of:
  * 6 PNE sessions (1 session of 90 minutes per week for 5 weeks).
  * 19 sessions of TE (2-3 weekly sessions of 60 minutes, for 7 weeks).
  Interventions: Behavioral: Pain Neuroscience Education (PNE)+ Therapeutic Exercise (TE)
- Usual treatment (Active Comparator): Delivery of a printed document with exercises to be performed at home for patients with persistent pain endorsed by a Scientific Society, as has been done in the Spanish Health Care Public System's usual practice with patients with chronic pain.
  Interventions: Behavioral: Active Comparator: Usual treatment

INTERVENTIONS:
Behavioral: Pain Neuroscience Education (PNE)+ Therapeutic Exercise (TE) — 12-week program consisting of PNE and TE
  Arms: Pain Neuroscience Education (PNE)+ Therapeutic Exercise (TE)
Behavioral: Active Comparator: Usual treatment — 12-week program consisting of home exercises, performed 3 days/week.
  Arms: Usual treatment

SUMMARY:
Justification: among the sequelae of Covid-19 in clinical practice we frequently find persistent neuromusculoskeletal pain. Previous studies carried out by this research group and in the scientific literature have shown that "Pain Neuroscience Education" (PNE) and Therapeutic Exercise (TE) constitute an effective care strategy in the treatment of persistent pain. Therefore, with this research we will try to respond with a treatment proposal from Primary Care (PC).

Objective: to determine whether an PNE and TE program is effective in patients presenting Long Covid Pain (LCP).

Method: Randomized clinical trial. A sample of 80 subjects will be recruited. The intervention group will receive a program of TE and PNE, of 12 weeks duration: 5 weeks of PNE, of 1 weekly session of 90 minutes, and 7 weeks of TE, with a total of 19 sessions of 60 minutes duration. The control group will receive the usual treatment. An assessment will be made at the beginning and after the end of the intervention, where the following variables will be measured: quality of life, intensity, distribution and expansion of pain, healthy physical condition and blood test values. These will be evaluated by means of physical examination, questionnaires and laboratory tests.

Applicability of the expected results: The proposed intervention is simple and reproducible. It requires few resources, and can produce changes in pain perception, functionality and quality of life in patients with LCP.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had Covid-19, with a confirmatory PCR+ test or positive antigen test and recorded in their primary care medical record.
* Subjects between 18-70 years old.
* Musculoskeletal pain of more than 12 weeks of evolution since the beginning of the infection.
* Agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* History of chronic musculoskeletal pain of more than 12 weeks of evolution prior to Covid-19.
* History of diagnosed major depression.
* Having a diagnosis of fibromyalgia prior to Covid-19 infection.
* Pregnancy.
* Pain of oncologic origin.
* Fracture or surgical intervention on the spine in the last year.
* Cognitive neurological impairment that prevents understanding of PNE contents (in case of doubt, assessment with Minimental state examination).
* Bladder or bowel incontinence.
* Saddle anesthesia.
* Patients with other clinical conditions that may aggravate chronic spine pain (chronic fatigue syndrome, fibromyalgia and complex regional pain syndrome).
* Patients with associated pathologies that make it impossible for them to perform TE.
* Patients undergoing treatment with alternative therapies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) | 3 months
  EQ-5D questionnaire (Quality of life 5 dimension questionnaire): The EQ-5D is a brief multi-attribute health status measure composed of five questions with Likert response options (descriptive system) and a visual analogue scale (EQ-VAS). The descriptive system covers five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with three levels of severity in each dimension (no problems, some problems, and extreme problems).

SECONDARY OUTCOMES:
Pain Intensity | 3 months
  Visual Analog Scale, VAS (0-100mm).
Body Chart | 3 months
  Nordic Questionnaire
Quantitative sensory tests | 3 months
  pain detection to pressure
Handgrip Strength assessment | 3 months
  With a manual dynamometer.
30 sit to stand test | 3 months
6 Minute Walking Test (6MWT) | 3 months
Maximal Inspiratory and Expiration Pressure (MIP/MEP) | 3 months
Catastrophism | 3 months
  Pain Catastrophism Scale (ECD).
Anxiety | 3 months
  Beck Anxiety Questionnaire (BAI)
Depression | 3 months
  Beck Depression Questionnaire-II (BDI-II)
Drug consumption. | 3 months
  Record by dose of the consumption of drugs for the patient's pain pre-post intervention.
Fatigue | 3 months
  Modified Fatigue Impact Scale (MFIS)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Valladolid, Valladolid, VALLADOLID, Spain

IPD SHARING:
Plan to Share IPD: No